CLINICAL TRIAL: NCT02707341
Title: CorEvitas Psoriasis (PSO) Registry
Brief Title: The CorEvitas Psoriasis (PSO) Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-PSO-500
Record Dates: First submitted 2015-05-04; First posted 2016-03-14 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis
Keywords: psoriasis; disease registry
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Psoriasis: Pts presenting to enrolling sites across the US are invited to enroll if eligible

SUMMARY:
The primary objective of the CorEvitas Psoriasis Registry is to study the comparative safety of approved psoriasis therapies in a North American cohort of psoriasis subjects treated by dermatologists. This includes assessing the incidence and nature of adverse events of special interest, including malignancy, in a real world population of psoriasis patients on new biologic therapies (e.g. secukinumab). Secondary objectives include analyzing the epidemiology and natural history of the disease, comorbidities, current treatment practices, and comparative effectiveness.

DETAILED DESCRIPTION:
Based on the operating procedures established by the Corrona Rheumatoid Arthritis (RA) Registry, the Psoriasis Registry will use a parallel structure based on a design and strategy developed by Corrona, LLC. This registry will be cooperatively managed by scientific, operational, and quality leaders at Corrona and medical leaders appointed by the National Psoriasis Foundation (NPF).

Investigators may enroll patients who have started on or switched to a systemic agent for psoriasis within the previous twelve months. Currently approved subcutaneous biologics are indicated for adult patients with chronic moderate to severe plaque psoriasis who are candidates for systemic therapy or phototherapy. The currently approved intravenous biologic agent is indicated for adult patients with chronic severe plaque psoriasis who are candidates for systemic therapy, and when other systemic therapies are medically less appropriate. All patients will receive standard of care treatments prescribed by the investigator, in accordance with the FDA-approved drug labeling, and all treatment decisions are the sole responsibility of the investigator.

This study will be conducted at approximately 200 sites across North America. Sites are assessed and selected through interviews with potential investigators and a corresponding site feasibility survey that includes information on the investigator's qualifications, previous research experience, and the availability of support staff, sub-investigators, and patient population.

The Corrona Psoriasis Registry is a longitudinal, observational study; therefore, the duration is indefinite with no pre-determined stop date. The enrollment period is estimated to take approximately four years, and subjects will be followed for a minimum of eight years beginning from the time the subject is enrolled.

The design is a prospective, multicenter, observational registry for subjects with psoriasis. Longitudinal follow-up data is obtained via Corrona Questionnaires completed by both subjects and their treating dermatologists (also known as "Providers" for a Corrona registry study) every 6 months (+/- 30 days). The registry is designed to collect data on patient demographics, smoking history, disease duration, disease severity, disease activity, history of prior psoriasis treatment, comorbidities, hospitalizations, adverse events of special interest, medication use, and laboratory results.

The registry is linked to external data sources including the Centers for Disease Control's National Death Index (NDI), the Centers for Medicare and Medicaid Services (CMS), and other administrative data sources to support drug safety monitoring and other research activities.

Any adverse events that are spontaneously volunteered by the subject or discovered as a result of general questioning by the investigator should be recorded on the Provider Follow-up Questionnaire for that visit.

ELIGIBILITY:
ELIGIBILITY CRITERIA∗ To be eligible for enrollment into the CorEvitas Psoriasis Registry, a patient must satisfy all of the inclusion criteria and none of the exclusion criteria listed below.

Inclusion Criteria:

The patient must:

1. Have been diagnosed with psoriasis by a dermatologist.
2. Be at least 18 years of age or older.
3. Be willing and able to provide written consent for participation in the registry.
4. Be willing and able to provide Personally Identifiable Information (PII) that includes the following types of personal information at a minimum: 1) Full Name and 2) Date of Birth.
5. Meet one of the following criteria.

Have started on or switched to a systemic psoriasis treatment within the previous 12 months†▲:

Exclusion Criteria:

1. Patient is participating in or planning to participate in a double-blind randomized of a psoriasis drug. Of note, concurrent participation in another observational registry or open-label Phase 3b/4 trial is not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled in the Psoriasis Registry during regularly-scheduled office visits. Selected dermatologists are invited to participate as investigators in the Registry. Physicians are selected carefully in an effort to ensure enrollment of subjects that represent a reasonable representation of a cross-section of the population throughout North America with Psoriasis. All potential sites are screened for clinical research experience and adherence to Good Clinical Practice (GCP) guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-04; Primary Completion 2100-12 (Estimated); Study Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs) or serious adverse events (SAEs). | A minimum of 8 years from last patient enrolled
  Targeted events include malignancy, cardiovascular disease, serious infection, inflammatory bowel disease, gastrointestinal perforation, neurological events, hepatic events, and general serious adverse events.
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Disease burden: Psoriatic area and severity index (PASI) | every 6 months for 8 years
Disease burden: Investigators Global Assessment (IGA) | every 6 months for 8 years
Disease burden: Body surface area (BSA) | every 6 months for 8 years
Percentage of patients with history of comorbidities | time frame: at registry enrollment
Physician reported: Fitzpatrick skin type | time frame: every 6 months for 8 years
Patient reported: EuroQOL-5D-3L | time frame: every 6 months for 8 years
Patient reported: Dermatology Quality of Life index (DLQI) | time frame: every 6 months for 8 years
Patient reported: Work productivity and Activity Impairment (WPAI) | time frame: every 6 months for 8 years
Patient reported: Pain, Fatigue, Itch score on Visual Analog Scale (VAS) (1-100) | time frame: every 6 months for 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Greenberg, MD, MPH, Study Director — CorEvitas

REFERENCES:
- [Derived] Armstrong AW, Feldman SR, Fitzgerald T, Alkousakis T, Sima A, Li A, Kang HJ, Main SI, Khattri S, Stein Gold L. Patient-Reported Outcomes by Baseline Body Surface Area Involvement Among Individuals Initiating Biologic Therapy: Results from the CorEvitas Psoriasis Registry. Dermatol Ther (Heidelb). 2025 Aug;15(8):2117-2130. doi: 10.1007/s13555-025-01456-5. Epub 2025 Jun 11. PMID 40498388
- [Derived] Strober B, Zhong Y, Sima A, Beeghly A, Eckmann T, Balagula E, Zhuo J, Lebwohl M. Criteria for Identifying Candidates for Systemic Psoriasis Treatment in the Real World: Application of the International Psoriasis Council Guidelines in Patients in North America. J Psoriasis Psoriatic Arthritis. 2024 Nov 21:24755303241302070. doi: 10.1177/24755303241302070. Online ahead of print. PMID 39583219
- [Derived] McLean RR, Sima AP, Beaty S, Jones EA, Eckmann T, Low R, McClung L, Spitzer RL, Stark J, Armstrong A. Durability of Near-Complete Skin Clearance in Patients with Psoriasis Using Systemic Biologic Therapies: Real-World Evidence from the CorEvitas Psoriasis Registry. Dermatol Ther (Heidelb). 2023 Nov;13(11):2753-2768. doi: 10.1007/s13555-023-01028-5. Epub 2023 Sep 27. PMID 37759099
- [Derived] McLean RR, Sima AP, Beaty S, Low R, Spitzer RL, Stark JL, Lesser E, Lee E, Armstrong A. Skin Clearance is Associated with Reduced Treatment Failure in Patients with Psoriasis: Real-World Evidence from the CorEvitas Psoriasis Registry. Dermatol Ther (Heidelb). 2023 Nov;13(11):2739-2751. doi: 10.1007/s13555-023-01027-6. Epub 2023 Sep 27. PMID 37755689
- See also: CorEvitas home page — https://www.corevitas.com/